CLINICAL TRIAL: NCT04585711
Title: Pharmacokinetics and Pharmacodynamics of Biologic Drugs in Obese Patients With Arthritis
Acronym: PRECISE
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: Funding expired
Sponsor: Duke University (Other)
Collaborators: National Institute of Arthritis and Musculoskeletal and Skin Diseases (NIAMS) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: Pro00105975; 1K23AR075874-01A1 (NIH)
Record Dates: First submitted 2020-10-07; First posted 2020-10-14 (Actual); Last update posted 2025-09-25 (Actual); Status verified 2025-09

CONDITIONS: Juvenile Idiopathic Arthritis; Rheumatoid Arthritis; Obesity
Keywords: Etanercept; Pharmacokinetics; Pharmacodynamics
MeSH Terms: conditions — Arthritis, Juvenile; Arthritis, Rheumatoid; Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Optimal dosing (Other): Obese children (≥ 2 year old) and adults with juvenile idiopathic arthritis (JIA) or Rheumatoid Arthritis (RA) who are starting etanercept as part of their routine medical care.
  Interventions: Drug: Etanercept Optimal dosing

INTERVENTIONS:
Drug: Etanercept Optimal dosing — Patients will receive Etanercept on an optimal dose interval over a 6-week period based on a PK/PD model.

SUMMARY:
The purpose of this study is to learn more about how adult and children's bodies use etanercept and how bodyweight influences how well etanercept works. This study will help us understand the proper dose of etanercept in obese children and adults.

DETAILED DESCRIPTION:
PRECISE is an open-label, single arm, single-center site study to evaluate the pharmacokinetics (PK) and pharmacodynamics (PD) of dosing interval-optimized etanercept in obese patients with Rheumatoid Arthritis (RA) and Juvenile Idiopathic Arthritis (JIA). Approximately 30 patients with JIA or RA who are starting etanercept standard-of-care will take part in the study.

Eligible patients will have blood collections before and after starting the biologic of interest to assess PK and disease activity. Five (5) blood samples will be collected through a combination of clinic and home visits.

ELIGIBILITY:
Inclusion Criteria

* Diagnosis of Rheumatoid Arthritis (RA) according to the 2010 American College of Rheumatology Classification Criteria (patients greater than or equal to 16 years of age at screening)
* Diagnosis of Juvenile Idiopathic Arthritis (JIA) according to the International League Against Rheumatism Classification Criteria (children less than 16 years of age at screening)
* Initiating treatment with etanercept as standard of care by a patient's primary rheumatologist
* Obese at baseline, defined as a body mass index (BMI) greater than or equal to 30 kg/m2 in subjects greater than or equal to 18 years of age, and a BMI greater than or equal to 95th percentile for age and sex in subjects less than18 years of age
* Active disease at screening, defined as a DAS28 > 3.2 in adults and JADAS27 > 3.8 in children
* Patients using oral corticosteroids (<10 mg) or DMARDs must be on a stable dose for at least 4 weeks prior to screening

Exclusion Criteria

* Receipt of any investigational medical product within the past 12 months
* Positive urine pregnancy test at screening or planned pregnancy during the study period
* Prior exposure to etanercept or any other biologic agent within 5 drug half-lives
* Contraindication to etanercept (e.g., allergy, current or chronic infection [positive tuberculosis screening test, positive hepatitis B surface antigen, positive hepatitis C antibody])
* Personal history of ever having malignancy, lymphoproliferative disease, or demyelinating disease
* Screening safety labs with a hemoglobin of ≤ 9 g/dL, white blood cell count <3.0x109L, platelets <125,000 x109L, AST/ALT more than 2x the upper limit of normal, or creatinine > 2 mg/dL for adults and >1 mg/dL for children
* Evidence of erosive osteoarthritis on plain films (if available at time of screening), or severe osteoarthritis (defined as any anticipated need for joint replacement within the next year) as judged by the primary rheumatologist
* History of any opportunistic infections, or recent severe infection in the 3 months prior to screening (e.g., hepatitis, pneumonia, pyelonephritis, bacteremia)
* Heart failure with NYHA classification 3 or more
* Severe functional impairment status, defined as HAQ >2 and CHAQ >1.75

Ages: 2 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2026-07-01 (Estimated); Primary Completion 2027-02-28 (Estimated); Study Completion 2027-02-28 (Estimated)

PRIMARY OUTCOMES:
Clearance (CL) | 6 weeks
  Clearance at steady state as measured by PK sampling
Volume of distribution (V) | 6 weeks
  Volume of distribution at steady state as measured by PK sampling

SECONDARY OUTCOMES:
Median prediction error between observed and model predicted concentrations | 6 weeks
  We will use PK/PD models to simulate drug concentration for each individual subject. We measure the error between simulated and observed plasma concentrations.
mean change in DAS28/JADAS27 | Baseline, 6 weeks
  We will score disease activity using the DAS28 (RA) or JADAS27 (JIA) at baseline and 6 week follow up. We will measure the change in score over 6 weeks.

CONTACTS AND LOCATIONS:
Overall Officials: Stephen Balevic, MD, Principal Investigator — Duke Clinical Research Institute
Locations (1):
- Duke University Medical Center, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No